CLINICAL TRIAL: NCT06718595
Title: Evaluation of Percutaneous Drainage of Appendicular Abscess, is There Any Need for Further Open Drainage ?
Brief Title: Study of Management of Appendicular Abscess
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, David Mamdouh Thabet, doctor, Assiut University
Other Study IDs: Appendicular abscess drainage
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Appendiceal Abscess

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to detect indications of surgical drainage after failure Ultrasound guided percutaneous drainage This study will include any male and female above 18 years old that presented with appendicular abscess Patients with appendicular abscess above the age of 18 years old All patients with generalized peritonitis or immunocompromised patients will be excluded from the study

DETAILED DESCRIPTION:
Prospective randomized study we will collect 30 patients diagnosed with appendicular abscess and they all will undergo Ultrasound guided percutaneous drainage of abscess and the group who will fail to insert the pigtail will undergo surgical drainage we will record the time of operation, number of cases with intraoperative complications and then follow up these patients during time of hospital stay for post operative pain and paralytic ileus

Study outcomes:

Primary outcomes:

1. Incidence of intra operative complications
2. Length of operations
3. Post operative pain
4. Incidence of intraoperative complications as injury of important structures
5. Lenght of hospital stay
6. Incidence of post operative complications related to surgery as wound infection, recurrence, intestinal obstruction

Secondary outcomes:

1. Cosmotic outcomes
2. Incidence of recurrence of pathology
3. Patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Patients with appendicular abscess above the age of 18 years old

Exclusion Criteria:

* Generalized peritonitis and patients with signs of spreading infection, toxemia and septicemia Multi-locular appendicular abscess Immunocompromised patients, hepatic dysfunction, renal impairment, uncontrolled patients and cardiac disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 100 patients was diagnosed with appendicular abscess in the emergency unit, department of general surgery, faculty of medicine, Assiut university
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
1-Incidence of intraoperative complications | Baseline

REFERENCES:
- [Background] Brown C, Kang L, Kim ST. Percutaneous drainage of abdominal and pelvic abscesses in children. Semin Intervent Radiol. 2012 Dec;29(4):286-94. doi: 10.1055/s-0032-1330062. PMID 24293801
- [Background] Darwazeh G, Cunningham SC, Kowdley GC. A Systematic Review of Perforated Appendicitis and Phlegmon: Interval Appendectomy or Wait-and-See? Am Surg. 2016 Jan;82(1):11-5. PMID 26802841
- [Background] Tannoury J, Abboud B. Treatment options of inflammatory appendiceal masses in adults. World J Gastroenterol. 2013 Jul 7;19(25):3942-50. doi: 10.3748/wjg.v19.i25.3942. PMID 23840138
- [Background] Deelder JD, Richir MC, Schoorl T, Schreurs WH. How to treat an appendiceal inflammatory mass: operatively or nonoperatively? J Gastrointest Surg. 2014 Apr;18(4):641-5. doi: 10.1007/s11605-014-2460-1. Epub 2014 Feb 4. PMID 24493295
- [Background] Bal A, Ozkececi ZT, Turkoglu O, Ozsoy M, Celep RB, Yilmaz S, Arikan Y. Demographic characteristics and seasonal variations of acute appendicitis. Ann Ital Chir. 2015;86:539-44. PMID 26899348